CLINICAL TRIAL: NCT00941174
Title: Folate Absorption Across the Large Intestine, Study #2: Capsule Study
Brief Title: Folate Absorption Across the Large Intestine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of Florida (Other)
Responsible Party: Principal Investigator, Deborah O'Connor, Associate Chief, Clinical Dietetics, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000008487-2b
Record Dates: First submitted 2009-07-14; First posted 2009-07-17 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: (13C5) Calcium Leucovorin; Folate absorption across the large intestine; Folate Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsule: 400 microg 13C5-Calcium-L-Leucovorin (Active Comparator)
  Interventions: Drug: 13C5-Calcium-L-Leucovorin
- IV Injection: : 100 microg 13C5-Calcium-L-Leucovorin (Active Comparator)
  Interventions: Drug: 13C5-Calcium-L-Leucovorin

INTERVENTIONS:
Drug: 13C5-Calcium-L-Leucovorin — This drug will be used in a clinical trial the objective of which is to determine whether, and to what extent, a physiological concentration of natural folate is absorbed across the large intestine with an intact microflora.
  Other Names: 13C5 Folate

SUMMARY:
The objective of this study is to determine whether the intact human colon with an unaltered microflora distribution absorbs folate and to what extent it is absorbed into the systemic circulation using a dual/oral intravenous route. This will elicit an understanding of colonic folate absorption and metabolism.

DETAILED DESCRIPTION:
This study supplements two earlier in print exploratory studies investigating the absorption of folate across the colon after an infusion during colonoscopy and a pre-trial with the purpose of determining dissolution characteristics of two placebo caplet formulations. Using a dual route oral/intravenous, folate (pharmaceutical name Calcium Leucovorin), labeled with a stable isotope will be used to quantitatively measure total folate levels, as well as the uptake of (13C) labeled folate. A pH dependent caplet targeted to the colon and fluoroscopy will determine dissolution characteristics. Labeled and unlabelled folate in blood and urine samples will be used to quantitatively measure the uptake of folate. This will further our understanding of the kinetics (caplet transit times), colonic folate absorption (metabolism) and impact on folate status (bioavailability) in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults
2. Age 18-65 years

Exclusion Criteria

1. <18 years of age, >65 years of age
2. chronic disease (eg. history of hepatic, gastrointestinal, renal, vascular, hematological, or neuropsychiatric disease) or surgery affecting gastrointestinal motility, pH or folate absorption/metabolism
3. regular use of medications affecting gastrointestinal pH, motility or folate absorption/metabolism (eg. anti-acid or nonsteroidal anti-inflammatory drugs [NSAIDS] such as aspirin/ibuprofen, phenytoin, sulfasalazine, phenobarbital, primidone, and cimetidine)
4. regularly consume > 1 drink of alcohol/d or current smoking (last 6 months)
5. planning a pregnancy, pregnant, breast feeding or the use of high-dose oral contraceptives/hormone replacement therapy
6. known sensitivity to Calcium Leucovorin
7. 130mL of blood is > 5% of total blood volume

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Blood Folate - Study Period 1 | Day 1 (Baseline), Day 2 (0h,1h,2h,3h,4h,5h,6h,7h,8h,9h,10h,11h,12h,24hr,48hr)
Blood Folate - Study Period 2 | Day 2 (0h, 0.25h,0.5h,1h,1.5h,2h,2.5h,3h,3.5h,4h)
Urine Folate - Study Period 1 | 24h, 48h, 72h, 96h
Urine Folate - Study Period 2 | 24h, 48h, 72h

SECONDARY OUTCOMES:
Dietary Recall Records for folate analysis during urine collection days, Anthropometric. | Study Phase 1 (Day 2,Day 3,Day 4,Day 5) Study Period (Day 2,Day 3,Day 4)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah O'Connor, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital For Sick Chidlren, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lakoff A, Fazili Z, Aufreiter S, Pfeiffer CM, Connolly B, Gregory JF 3rd, Pencharz PB, O'Connor DL. Folate is absorbed across the human colon: evidence by using enteric-coated caplets containing 13C-labeled [6S]-5-formyltetrahydrofolate. Am J Clin Nutr. 2014 Nov;100(5):1278-86. doi: 10.3945/ajcn.114.091785. Epub 2014 Sep 3. PMID 25332326